CLINICAL TRIAL: NCT01476748
Title: A Pilot Study to Determine the Extent of Intraoperative Laparoscopic Trocar Slippage.
Brief Title: Intraoperative Trocar Slippage Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jon I. Einarsson, MD, MPH, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2011P001825
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Trocar Slippage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ethicon Xcel Trocars (Active Comparator): Ethicon Xcel trocars will be used in this arm with Laprostop device
  Interventions: Device: LaproStop
- Covidien Veraport Trocars (Active Comparator): Covidien Veraport Trocars will be used in this arm with the Laprostop device
  Interventions: Device: LaproStop
- Storz Reusable Trocars (Active Comparator): Storz Reusable Trocars will be used in this arm with the Laprostop device
  Interventions: Device: LaproStop

INTERVENTIONS:
Device: LaproStop — One of the subject's trocars will be randomized to be used with a LaproStop device.

SUMMARY:
The purpose of this study is to find out how much a trocar might slide during a typical laparoscopic hysterectomy. We also want to find out if there is a difference between how much three commonly used trocars slide and if a device called LaproStop has an effect on the slippage.

Patients will be randomly assigned into the different trocar groups. After this assignment has been made, we will then assign the Laprostop to one of the two trocars by chance.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a hysterectomy at Brigham and Women's Hospital and Faulkner Hospital.

Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon I Einarsson, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Minimal Invasieve Gynaecology Surgery, Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in a tertiary hospital, from 12-26-12 to 06-18-13
Pre-assignment Details: All enrolled participants were included in the trial
Groups:
- Covidien Veraport Trocars; Ethicon Xcel Trocars; Storz Reusable Trocars: LaproStop : One of the subject's trocars will be randomized to be used with a LaproStop device.
Period: Overall Study
Arm/Group | Covidien Veraport Trocars | Ethicon Xcel Trocars | Storz Reusable Trocars
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Covidien Veraport Trocars | Ethicon Xcel Trocars | Storz Reusable Trocars | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 15
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (2.48) | 43 (9.61) | 44.6 (6.34) | 45.13 (6.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 15
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Secondary Outcome: Trocar Slippages Without LaproStop
Description: Number of participants with slippages with LaproStop
Time Frame: During the hysterectomy procedure, up to 2 hours and 32 minutes
Measure: Number; unit: Participants
Groups:
- Covidien Versaport Trocars; Ethicon Xcel Trocars; Storz Reusable Trocars: LaproStop : One of the subject's trocars will be randomized to be used with a LaproStop device.
Arm/Group | Covidien Versaport Trocars | Ethicon Xcel Trocars | Storz Reusable Trocars
Number analyzed (Participants) | 5 | 5 | 5
Participants | 0 (4.47) | 2 (2.68) | 4 (2.4)

2. Primary Outcome: Trocar Slippages With LaproStop
Description: Number of participants with slippages with LaproStop
Time Frame: During the hysterectomy procedure, up to 2 hours and 32 minutes
Population: Pilot study
Measure: Number; unit: Participants
Arm/Group | Covidien Versaport Trocars | Ethicon Xcel Trocars | Storz Reusable Trocars
Number analyzed (Participants) | 5 | 5 | 5
Participants | 1 | 2 | 3

ADVERSE EVENTS:
Arm/Group | Covidien Veraport Trocars | Ethicon Xcel Trocars | Storz Reusable Trocars
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
There were no adverse events encountered during this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes